# Exploring Uterine Cancer Clinical Trials - Revealing Participation Patterns in Individuals With Uterine Cancer

Navigating the Informed Consent Procedure within <u>Power Clinical</u> <u>Trial's</u> Observational Study: An Informative Document for Uterine Cancer Patients

Date: August 11, 2023

Understanding the Essence of This Informed Consent Form

If you're tasked with completing this form, it signifies your possible participation in an observational clinical trial specifically designed for individuals navigating uterine cancer. This form acts as an extensive guide, revealing the study's overarching objectives, meticulous execution plan, and diverse implications, both advantageous and potentially otherwise. Taking the time to thoughtfully contemplate your potential involvement before making a decision is crucial, and seeking guidance from a trusted confidant can offer valuable insights. If any intricacies of the information enclosed within this document remain unclear or if questions arise, rest assured that the researcher is prepared to offer clarifications.

## Study Focus

Uterine cancer, also known as endometrial cancer, is a type of cancer that originates in the lining of the uterus, which is called the endometrium. The uterus is a female reproductive organ where a fertilized egg implants and develops into a fetus during pregnancy.

In uterine cancer, the cells of the endometrium undergo abnormal growth and multiplication, forming a tumor. This tumor can be benign (not cancerous) or malignant

(cancerous). Malignant uterine tumors have the potential to invade nearby tissues and spread to other parts of the body, a process known as metastasis.

Clinical trials targeting uterine cancer play a pivotal role in assessing the safety and efficacy of emerging treatments for this condition. These trials are pivotal in determining whether these novel treatments outshine existing options and offering robust evidence to endorse their broader application.

This study primarily delves into examining the experiences of individuals diagnosed with uterine cancer as they actively participate in a distinctive clinical trial encompassing medical interventions. The central focus revolves around meticulously tracking trial completion rates and instances of voluntary withdrawal among these participants.

#### Introduction to Observational Studies

As a participant in this medical trial, you will be taking part in an observational study, a specific type of clinical trial designed to gather information by observing individuals without introducing any changes to their care plans.

Researchers will simply observe your progress and assess the outcomes of your condition without making any interventions. This kind of trial plays a crucial role in deepening our understanding of the natural progression of a specific condition and its impact on individuals who have been diagnosed with it. By participating in this observational study, you will play a valuable role in advancing medical knowledge and contributing to the enhancement of care for individuals sharing the same condition.

# Insights into Upcoming Uterine Cancer Clinical Trials

It's important to recognize that this clinical trial employs an observational approach, meaning that your participation will not involve the application of specific treatments or interventions as part of the study. However, the realm of uterine cancer clinical trials encompasses a spectrum of variations, including interventional trials that require participants to undergo particular treatment protocols.

Making a well-informed decision about your potential involvement in a clinical trial calls for a proactive approach to researching and comparing various studies. An abundance of information regarding <u>uterine cancer-related trials</u> can be accessed through platforms like clinicaltrials.gov. Additionally, Power's dedicated website showcases a range of

ongoing <u>uterine cancer clinical trials</u> actively seeking participants. By investing time in thorough research and understanding the diverse array of clinical trial formats, you can confidently make a decision about your participation in a trial.

#### Participation by Choice in Clinical Trial Surveys

As a participant in this observational clinical trial, we extend an invitation to share your unique experiences with us. This will entail the completion of questionnaires every two weeks, with an estimated time commitment of around 20-30 minutes. Furthermore, on a quarterly basis, we will arrange check-in calls for the duration of your active involvement in the trial.

It's imperative to underscore that your participation in the survey component of the trial is entirely voluntary. You have the autonomy to decide whether to respond to specific questions or all questions, and you hold the right to discontinue your participation in the trial whenever you deem fit. We acknowledge that the decision to engage in a clinical trial is deeply personal, and our commitment is to offer unwavering support throughout your journey. Your privacy and comfort hold the highest priority, and we are dedicated to honoring your decision-making process throughout the trial.

## Preserving the Privacy of Your Replies

Safeguarding the confidentiality of your information is a fundamental principle throughout the entire span of this clinical trial. In order to maintain your anonymity, we kindly urge you not to disclose any personal or identifiable particulars in your responses to the questionnaires. The dedicated research team is fully devoted to reinforcing the protective veil of your privacy. However, it's important to note that specific legal situations may arise, mandating the release of your data.

# Possible Advantages

While immediate benefits might not be immediately apparent to individuals taking part in this observational clinical trial, their involvement holds the potential to create a lasting impact on the lives of others. The reservoir of data collected from participants will contribute to refining future procedures for enrolling uterine cancer patients, ultimately leading to greater access to medical research opportunities. By embarking on this

clinical journey, individuals have the chance to become agents of transformative change in the field of medical research, significantly influencing the trajectory of future uterine cancer patients.

#### Potential Hazards

The realm of clinical trials has unquestionably propelled medical advancement, yet it is equally important to acknowledge the potential specter of health risks that can hang over participants, especially in trials involving novel treatments.

However, our observational clinical trial stands apart, effectively mitigating this risk by avoiding the requirement for participants to undergo new interventions. Instead, the central focus is on observation and outcome measurement, without introducing any unwarranted health hazards.

Embarking on a Deeper Exploration of Inclusivity in Clinical Trials

For those who harbor an interest in delving into the intricate landscape of representation within clinical trials, an array of online resources stands ready for your enthusiastic engagement.

Whether you aim to decipher the intricacies interwoven with challenges and prospects, or simply seek to enhance your personal voyage through the realm of clinical trials, these reservoirs of knowledge shine as illuminating sources:

Goodson, Noah, Paul Wicks, Jayne Morgan, Leen Hashem, Sinéad Callinan, and John Reites. "Opportunities and counterintuitive challenges for decentralized clinical trials to broaden participant inclusion." *NPJ Digital Medicine* 5, no. 1 (2022): 58.

<u>Dalton, Emily J., Natasha A. Lannin, Bruce CV Campbell, Leonid Churilov, and Kathryn S. Hayward. "Enhancing generalizability of stroke clinical trial results: Illustrations from upper-limb motor recovery trials." *International Journal of Stroke* 18, no. 5 (2023): 532-542.</u>

Confirmation of Informed Agreement

I hereby affirm that I have dedicated substantial time to comprehensively understand and assimilate the contents encapsulated within the informed consent form, either independently or with the support of a trusted individual who has conveyed its essence to me. All inquiries and reservations that occupied my thoughts have been diligently addressed to my utmost satisfaction.

I am fully cognizant that my involvement in this study arises from a voluntary choice, and the authority to retract my consent resides solely with me, without any obligation to provide a rationale or face financial obligations. It has been explicitly communicated to me that a duplicate of this informed consent form will be provided for my archival purposes.

Having meticulously considered and evaluated the entirety of the information presented to me, I hereby express my concurrence to partake in this study, a reflection of my independent volition.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| <br>Date |

Validation by Informed Consent Facilitator

I confidently confirm that I have engaged in a thorough dialogue with the participant, carefully unraveling the complexities enshrined within this textual document. My aim was to ensure the participant's comprehensive understanding of the trial's overarching objectives, employed methodologies, potential risks and benefits, as well as other vital components intrinsic to the uterine cancer clinical trial.

Adequate space was afforded to the participant, encouraging the emergence of inquiries and facilitating the clarification of uncertainties or misconceptions. It is of utmost importance to highlight that the participant's involvement in this trial is a result of their voluntary choice, and they possess the unrestricted right to discontinue their participation at any point, driven by any reason, without bearing any financial obligations.

Upon the participant's provision of consent, a meticulously preserved duplicate of this textual document was provided to them, serving as a repository for their personal records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| Date. |